CLINICAL TRIAL: NCT02695251
Title: Renal Hemodynamic, Functional and Metabolic Changes After AGEs (Advanced Glycation End Products) Load by Positron Emission Tomography (PET) and Blood Oxygen Level-Dependent (BOLD) - MRI. The AGE- Functional Reserve Study.
Brief Title: AGE - Functional Reserve
Acronym: AGE-FR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 69HCL15_0122
Record Dates: First submitted 2016-02-26; First posted 2016-03-01 (Estimated); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Kidney Function Tests

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low AGE meal (Experimental): Renal functional parameters are measured at baseline and after a low AGE (eggs) meal
  Interventions: Other: low AGE meal
- High AGE meal (Experimental): Renal functional parameters are measured at baseline and after a high (mixed nuggets) AGE (eggs) meal
  Interventions: Other: High AGE meal

INTERVENTIONS:
Other: low AGE meal — Patients will receive a low AGE (eggs) meal
  Arms: Low AGE meal
Other: High AGE meal — Patients will receive a high (mixed nuggets) AGE (eggs) meal
  Arms: High AGE meal

SUMMARY:
Renal functional reserve is defined as the glomerular hyper filtration induced by a protein load. Renal blood flow and Glomerular Filtration Rate (GFR) increase in response to a protein load. Renal functional reserve loss is associated with a persistent hyper filtration state, seen in first stages of diabetic nephropathy, leading to progression of Chronic Kidney Disease (CKD). This observation has lead to larger clinical studies that demonstrated the positive effects of protein restriction on kidney function, and allowed the scientific community to recommend low proteins diet (less than 0.8 g / kg/ day) to prevent CKD progression. Nevertheless, the precise mechanisms responsible for kidney hemodynamic and metabolic changes induced by a protein load, are debated. Uribarri et al have suggested that renal hemodynamic changes induced by a protein load are mainly due to the Advanced Glycation End Products (AGEs) content. Indeed, initial studies experimental conditions leading to the demonstration of renal functional reserve (amino acid or protein perfusion or cooked meat), were in fact responsible for an AGEs load, based on recent published data.

The aim of this study is to determine whether AGEs alone or proteins in general are responsible for the mobilization of renal functional reserve, leading to the progression of CKD.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males subjects
* age between 18 and 30 years old

Exclusion Criteria:

* Kidney disease
* Diabetes
* Obesity
* Hypertension
* Non Steroidal Anti Inflammatory Drug treatment (NSAIDS)
* MRI Contra indications
* Myeloma
* High basal Radiation exposure : more than 1 milliSievert (mSv) in the last 6 months

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Renal Blood Flow | 120 minutes after meal
  Differences in Renal blood flow will be assessed 120 minutes after 2 different meals, either high AGE (mixed nuggets) or low AGE meal (mixed eggs), with PET- MRI using 150 labeled water.

SECONDARY OUTCOMES:
renal oxygen content | 120 minutes after meal
  Differences in renal oxygen content will be assessed after either a high or low AGE meal with BOLD (Blood Oxygen Level Dependant) - MRI
renal oxidative metabolism | 120 minutes after meal
  Differences in renal oxidative metabolism will be assessed after either a high or low AGE meal with PET MRI using 11C labeled - Acetate

CONTACTS AND LOCATIONS:
Overall Officials: Laurent JUILLARD, MD, PhD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Service de Néphrologie - Hôpital Edouard Herriot, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Normand G, Lemoine S, Villien M, Le Bars D, Merida I, Irace Z, Troalen T, Costes N, Juillard L. AGE Content of a Protein Load Is Responsible for Renal Performances: A Pilot Study. Diabetes Care. 2018 Jun;41(6):1292-1294. doi: 10.2337/dc18-0131. Epub 2018 Apr 2. PMID 29610272